CLINICAL TRIAL: NCT04932811
Title: The Lung Microbiome in Patients With Emphysema and Chronic Obstructive Lung Disease Treated With Endobronchial Valves: Complications and Prognosis
Brief Title: The Lung Microbiome and Endobronchial Valve Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Hermann, Cand. med., Aarhus University Hospital
Other Study IDs: 1-10-72-323-20
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fluid from bronchioalveolar lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung emphysema is often associated with chronic obstructive pulmonary disease (COPD) and without any cure. Dyspnea is the main, debilitating symptom and is relieved by inhaled bronchodilators and rehabilitation. However, a substantial number of patients continue to suffer from dyspnea and among these, many patients have severely hyperinflated lungs due to predominant emphysema. For selected patients, lung transplantation or lung volume reduction by surgical removal (LVRS) of the most emphysematous parts of the lung can improve symptoms and survival. However, LVRS is related to complications and not all patients are suitable for surgery. An alternative to LVRS is bronchial lung volume reduction with endobronchial valves (EBV). One-way valves are inserted in the bronchial system using a bronchoscope and it has emerged as a valid treatment option with similar effects as LVRS with reduction of hyperinflation and increasing pulmonary function, quality of life, and exercise capacity.

The normal lung is colonized with several types of bacteria, and together this is called the microbiome. Some bacteria are potentially beneficial, while others are potentially harmful. After the insertion EBV, some patients develop chronic infections. The hypothesis is that the microbiome can affect the risk of this chronic infection, and therefore the objective of this study is to access the microbiome during the insertion of the EBV, and afterwards observe which patients develop chronic infection and if these patients are harbouring specific types of bacteria.

DETAILED DESCRIPTION:
The objective of this study is primarily to investigate the significance of the lung microbiome on the outcome and morbidity after EBV treatment. Second, to investigate the evolution of the lung microbiome in patients later requiring valve removal or clean-up.

Before the insertion of the EBV, but during the procedure, the patient will undergo a bronchoalveolar lavage (BAL). BAL fluid will undergo bacterial profiling through S16-ribosomal analysis and ordinary bacterial culturing. Number of infections and need for clean-up or valve removal will be registered during the following 24 months, where the patient follows the ordinary follow-up programme. As a secondary part of the study, during the potential clean-up or valve removal, the removed material will again undergo S16-ribosomal analysis and bacterial culturing to investigate shift in microbiome.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with emphysema selected for EBV treatment by multidiciplinary team, independent of this study.
* Written informed consent

Exclusion Criteria:

- Intake of oral antibiotics within 1 month before the procedure. Patients receiving preventive long-term treatment with antibiotics can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with emphysema treated at Aarhus University Hospital, Odense University Hospital or Rigshospitalet, selected for EBV treatment independent from this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-16 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary infection | 2 years
  Number and severity of pulmonary infection after surgery
Valve dysfunction | 2 years
  Dysfunction of valves requiring clean up
Microbiome | During surgery
  Microbiome in bronchioalveolar lavage

SECONDARY OUTCOMES:
Formation of atelectasis | 2 years
  Formation and maintainance of atelectasis after insertion of valve

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No